CLINICAL TRIAL: NCT02803723
Title: "Holding-cuddling" Plus Oral Sucrose Versus Oral Sucrose for Reducing Venipuncture Pain in Newborns and Infants
Acronym: Casa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015/CHU/08
Record Dates: First submitted 2016-05-30; First posted 2016-06-17 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2016-05

CONDITIONS: Blood Sampling
MeSH Terms: interventions — Sucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Holding-cuddling + Sucrose (Experimental): The Holding-cuddling is started 5 minutes before and the sucrose administration is started 2 minutes before blood sampling.
  Interventions: Procedure: Holding-cuddling; Procedure: Sucrose
- Sucrose alone (Active Comparator): The sucrose administration is started 2 minutes before blood sampling.
  Interventions: Procedure: Sucrose

INTERVENTIONS:
Procedure: Holding-cuddling — The "Holding-cuddling" is started 5 minutes before veinipuncture.
  Arms: Holding-cuddling + Sucrose
Procedure: Sucrose — The sucrose adminstration is started 2 minutes before veinipuncture.

SUMMARY:
"Holding-cuddling" plus oral sucrose versus oral sucrose for reducing venipuncture pain in newborns and infants.

Neonates and infants routinely undergo venipuncture in pediatric and neonatal intensive care units.

Such procedure is painful and several units administer 24% oral sucrose with pacifier during venipuncture, as this non-pharmacological intervention is considered safe and effective for procedural pain relief in infants from birth to 3 months of age. However, several studies point out that further research is needed to assess its efficacy in combination with other behavioral interventions for analgesia during painful procedures. Current knowledge suggests that multisensorial stimulation associated with oral sucrose could allow even more effective analgesia. To date, the studied stimulation strategies are based on massage, voice, eye contact and fragrance during heel prick. The "holding-cuddling" - that is the fact of holding the child in a safe, reassuring and warm position during the examination or medical intervention is promoted by various hospitals in order to favor the comfort of all the caregivers during such a procedures. This intervention should be primarily parents-driven but, in case of unavailability, it can be performed by the nursing staff. The hypothesis of this study is that the combination of "holding-cuddling" plus oral sucrose in more effective than oral sucrose in diminishing behavioral pain response during a venipuncture in newborns or infants less than three-month-old.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization at CHU de la Réunion - site sud in Neonatal Intensive Care Unit or Neonatology Unit. (Neonate reanimation, pediatric reanimation or Neonatology services)
* Informed consent from holder(s) of the parental authority

Exclusion Criteria:

* Intubated ou sedated patients
* Treated with a combined analgesic during venipuncture
* Having indications against sucrose
* For which behavorial items from DAN scale are difficult to evaluate regarding their pathology (ex: severe neuromotor handicap)

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Evolution of Pain | At 0 and 30 seconds after the veinopuncture
  Measure of pain by DAN scale at the time of the veinopuncture

SECONDARY OUTCOMES:
Cardiac Frequency | At 0 and 30 seconds after veinopuncture
  Measure of the cardiac frequency at the time of the veinopuncture and 30 seconds after
Oxygen saturation | At 0 and 30 seconds after veinopuncture
  Measure of the oxygen saturation at the time of the veinopuncture and 30 seconds after
Pain at 1 min | 1 min after veinopincture
  Measure of pain by DAN scale 1 minute after veinopuncture

CONTACTS AND LOCATIONS:
Overall Officials: Francesco BONSANTE, MD, Principal Investigator — CHU de La Réunion; Silvia IACOBELLI, MD, Principal Investigator — CHU de La Réunion

IPD SHARING:
Plan to Share IPD: No